CLINICAL TRIAL: NCT03986788
Title: Effet de l'Impesanteur Sur la Distribution du débit Sanguin cérébral.
Brief Title: Cerebral Blood Flow Distribution During Parabolic Flight-induced Microgravity
Acronym: GraCer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Hospital, Caen (Other)
Collaborators: Centre National d'Etudes Spatiales (Other Government); Université de Caen Normandie (Other); The University of New South Wales (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-A01090-55
Record Dates: First submitted 2019-05-23; First posted 2019-06-14 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Weightlessness; Cerebral Blood Flow
MeSH Terms: interventions — Weightlessness

STUDY DESIGN:
Intervention Model Description: Comparison of cerebral blood flow in 1G, 1.8 G and 0G conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Weightlessness (Other): Weightlessness measurements during flight
  Interventions: Other: Weightlessness

INTERVENTIONS:
Other: Weightlessness — Volunteers will be studied during parabolic flight. Cerebral blood flow will be measured in different part of the brain during weightlessness ans compared to 1g and hypergravity measurements.

SUMMARY:
When astronauts return from space flight, they manifest a set of symptoms, the most striking of which is orthostatic intolerance, that is, the inability to stay upright. This orthostatic intolerance is related to cardiovascular adaptation and disappears in a few days, but the prospect of long-term space travel makes this maladaptation a major concern of space agencies, at a time when there is serious consideration to make " land "a ship on Mars.

Previous studies suggest that brain vessel adaptation may contribute to spatial post-flight orthostatic intolerance. The question remains controversial because not all studies are consistent. These studies are all based on the measurement of blood flow in a single artery of the brain (the average cerebral, see cerebral circulation diagram) easily accessible with a Doppler ultrasound machine. Our team has good reason to believe that the adaptation of the cerebral vessels is not carried out in the same way in all the arteries of the brain and that in particular the arteries that irrigate the posterior and inferior parts of the brain are a major determinant. from cerebrovascular adaptation to orthostatism and that orthostatic intolerance is more specifically related to a decrease in blood flow in these arteries. On the other hand our team has shown that the external carotid artery plays, under certain conditions, a buffer role of the sudden variations of perfusion pressure of the brain.

During the weightless phase of parabolic flight, part of the blood from the legs and abdomen "rises" to the thorax and this transfer of fluid induces changes in blood pressure and cardiac output that affect the cerebral circulation. From a cardiovascular point of view, it is the same thing for a seated subject to lie down, but the parabolic flight offers the unique possibility of achieving this transfer in a fraction of a second and thus allowing to study the immediate response of the cerebral circulation. .

Investigators goal is therefore to quantify the changes in blood flow in the posterior and anterior territories of the brain (transcranial ultrasound) as well as in the internal carotid and vertebral (Doppler ultrasound) during changes in blood pressure and cardiac output induced by transfers. liquid resources associated with the transition to weightlessness.

The oxidative stress generated by weightlessness has been identified as a determining factor in cerebrovascular deconditioning associated with orthostatic intolerance. In order to quantify the biochemical markers of this stress, a venous sample will be taken before and just after the parabolic flight.

DETAILED DESCRIPTION:
Parabolic flights make it possible to produce a reduced gravity environment on Earth. With the specially adapted A310 Zero-G, each parable produces a period of zero gravity ("0g"). The duration of the periods of reduced gravity is about 21 seconds. Each parable begins and ends with a resource (hyper-gravity) at 1.8 g; each resource lasts about 20 seconds. A typical flight lasts from two to three hours and includes 30 parabolic maneuvers, usually all in weightlessness.

Participants will arrive at Novespace, at Bordeaux-Mérignac Airport, no later than 2 pm the day before the first flight of the campaign in order to participate in the security briefing. A delay of at least 2 hours will be granted before collection of their written consent.

Before the flight, the participants will necessarily participate in the safety briefing (2h, organized by the Flight Manager (Novespace) and will meet the research team to become familiar with the procedures and devices that will be used during the experiment.

On the day of the flight, the participants will have to arrive at the premises of Novespace before 7.30am.

Before the flight, they will be prepared for flight recordings. Seven self-adhesive electrodes will be placed on the chest to measure the electrical activity of the heart and the blood volume in the chest.

A venous blood test to measure blood markers of oxidative stress will be performed by a doctor or a registered nurse.

Doppler and ultrasound operators will make blood flow measurements in the vertebral, internal carotid, posterior cerebral and anterior cerebral arteries) using an echo-doppler device. These measures are strictly non-invasive and painless. Participants can take medication against motion sickness under the supervision of the flight doctor. The duration of the study is a little less than 6 hours (2 hours before the flight, 3 hours flight, 30 minutes after the flight).

Preparation before parables, in the plane. In addition to the participant, two other subjects will be the participants of the flight, one will also be a subject, and the third will be a rescue participant who will be tested in case the subject or his partner falls ill during the flight. The flight includes 31 parables, but the first participant will be subject only for 16 parables and the second for 15.

When it is not subject, the participant is rid of equipment and can join the so-called "free floating" area to enjoy the sensations of weightlessness.

After takeoff, but before the first parable the subject (or the other participant) will sit on a chair built for the flight. His pelvis will be immobilized by restraints to prevent him from floating freely during the weightlessness.

It will be connected to different measuring equipment, all non-invasive:

An arterial pressure sensor on the finger. Electrotrocardiogram (connected to 3 self-adhesive electrodes) Thoracic impedance meter (connected to 4 self-adhesive electrodes) An oxygen scope (for measuring the expired CO2).

During the flight During each phase of weightlessness, an operator will apply on the neck or skull of the subject an ultrasound measurement probe (as on the ground). We recommend that participants do not move their head, especially during periods of hypergravity, to prevent motion sickness.

Except in exceptional circumstances, the aircraft normally completes the mission, but it must be clear that the subject is free to withdraw his consent and participation in the experiment at any time, without prejudice to him or to any other reason, without justification, including during the flight.

After the flight Following the flight, a second venous sample will be made to determine the effects of weightlessness on the markers of oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (men or women)
* Aged from 18 to 65
* Affiliated to a Social Security system and, for non-French resident, holding a European Health Insurance Card (EHIC)
* Who accepted to take part in the study
* Who have given their written stated consent
* Who have passed a medical examination similar to a standard aviation medical examination for private pilot aptitude (JAR FCL3 Class 2 medical examination). There will be no additional test performed for subject selection.

Exclusion Criteria:

* Persons who took part in a previous biomedical research protocol, of which exclusion period is not terminated.
* Persons with history of cerebral, cardiovascular or vestibular diseases.
* Pregnant women (urine pregnancy test for women of childbearing potential)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Cervical blood flow | baseline
  Measurement of the cervical blood flow in external (ECA), internal (ICA) and vertebral arteries (VA).
  ICA, VA and ECA blood flow velocities will be measured with a color-coded ultrasound system (Vivid-e; GE Healthcare, Tokyo, Japan) equipped with a 10 MHz linear transducer. ICA blood flow measurements will be performed 1.0-1.5 cm distal to the carotid bifurcation while the subject's chin will be slightly elevated. VA blood flow will be measured between the transverse processes of C3 and the subclavian artery. The systolic and diastolic diameters will be measured in detail, and then the mean diameter (in centimetres) will be calculated in relationship to the blood pressure curve, as follows: mean diameter = (systolic diameter×1/3) +(diastolic diameter × 2/3).
Transcranial blood flow | baseline
  Measurement of the transcranial blood flow in anterior (ACA), middle (MCA) and posterior (PCA) cerebral arteries. Blood flow velocities in PCA, MCA and ACA will be measured with an echo-doppler device (Philips CX50, Philips, the Netherlands) using vascular probes adapted to transcranial Doppler. Flows in the different branches of the circle of Willis (ACA-1, MCA-1, PCA-1, ACoA, PCoA) will be used to assess the cerebral hemodynamic indices.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Kassel, Hospital Manager, Study Director — University Hospital, Caen
Locations (1):
- Novespace A310-0G, Mérignac, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Site for weightlessness experimentations — http://www.novespace.fr/